CLINICAL TRIAL: NCT04514471
Title: Feasibility of Conducting a Telehealth Study Assessing the Removal of Filter Ventilation on Smoking Behavior and Biomarkers
Brief Title: Feasibility Study - Filter Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020LS110; NCT06439238 (obsolete NCT alias)
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: Open label, between-subject, randomized multi-center pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unventilated Filter Cigarette (Experimental): Conventional cigarette with approximately 6-7% (non-menthol) and 5-6% filter ventilation (menthol).
  Interventions: Other: Unventilated filter cigarettes
- Ventilated Filter Cigarette (Active Comparator): Conventional cigarette with approximately 22-26% (non-menthol) and 35-38% filter ventilation (menthol).
  Interventions: Other: Ventilated filter cigarettes

INTERVENTIONS:
Other: Unventilated filter cigarettes — Currently marketed unventilated cigarettes
  Arms: Unventilated Filter Cigarette
Other: Ventilated filter cigarettes — Currently marketed ventilated cigarettes
  Arms: Ventilated Filter Cigarette

SUMMARY:
This open label, between-subject, randomized multi-center pilot study will assess the feasibility of conducting a study remotely with telehealth visits to assess the effect of cigarettes with minimal filter ventilation vs. moderate filter ventilation on smoking behavior and biomarkers of tobacco toxicant exposure. Subjective measures, alveolar carbon monoxide, blood pressure and cigarettes per a day will be collected remotely. Biological samples will be collected at home and mailed to the study clinic.

DETAILED DESCRIPTION:
Smokers of cigarettes with about 16-30% ventilation in their conventional cigarettes who meet eligibility criteria will enter 3 weeks of monitoring of usual brand smoking. Subjects will then be randomly assigned for a period of 6 weeks to one of two conditions: 1) ventilated cigarettes; or 2) unventilated cigarettes. Subjects in each condition will be unblinded to simulate real world conditions. Subjects are provided with a debit card (ClinCard) that has been loaded with the appropriate amount of money to cover self-purchased usual brand cigarette in baseline and the assigned study cigarettes during intervention. Weekly telehealth visits will be conducted during baseline and the 6 weeks on study cigarettes to collect study measures, followed by a one month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Regular cigarette smoker
* Currently smoking an eligible brand
* Generally good health
* Access to smartphone or tablet and a device with a functioning camera for telehealth visits. Also must have internet access.

Exclusion Criteria:

* Unstable health
* Uncontrolled high blood pressure
* Pregnant or breast-feeding

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of approach - Drop outs | Baseline through Week 6
  Percent of drop-outs in baseline and post-randomization.
Feasibility of approach - Missing Data | Baseline through Week 6
  Extent (percent) of missing data
Feasibility of approach - Participant Satisfaction | Baseline through Week 6
  Degree of difficulty collecting data through telehealth visits, mailing in biosamples and self-purchase of cigarettes (descriptive statistics (e.g., percent or mean responses)

SECONDARY OUTCOMES:
Change in Total Nicotine Equivalents (TNE) | effect size for each arm calculated as the baseline minus the 6 week value divided by the SD of this difference
  The sum of nicotine and its metabolite concentrations used for evaluating nicotine exposure.
Change in 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) | effect size for each arm calculated as the baseline minus the 6 week value divided by the SD of this difference
  One of the tobacco specific nitrosamines, one of the most important groups of carcinogens in tobacco products, which are formed from nicotine during the curing and processing of tobacco.
Change in mean cigarettes per day (CPD) | effect size for each arm calculated as the baseline minus the 6 week value divided by the SD of this difference
  The change in mean cigarettes per day (CPD) based on 7 day ITR data before visit 00 and week 6 visit.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PH.D, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Undecided